CLINICAL TRIAL: NCT06188559
Title: An Open-label, Multicenter, Phase 2 Dose Optimization and Expansion Study to Evaluate the Safety and Efficacy of BB-1701, an Anti-human Epidermal Growth Factor Receptor 2 (Anti-HER2) Antibody-drug Conjugate (ADC), in Previously Treated Subjects With HER2-positive or HER2-low Unresectable or Metastatic Breast Cancer
Brief Title: A Study of BB-1701 in Previously Treated Participants With Human Epidermal Growth Factor Receptor 2 (HER2)-Positive or HER2-low Unresectable or Metastatic Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Collaborators: Bliss Biopharmaceutical (Hangzhou) Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BB-1701-G000-205; 2023-506866-30 (Other: EU-CT Number)
Record Dates: First submitted 2023-11-28; First posted 2024-01-03 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Breast carcinoma; Unresectable or metastatic breast cancer; HER2-positive or HER2-low unresectable or metastatic breast cancer; BB-1701
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: For Dose Optimization (Part 1), this study is randomized and for Dose Expansion (Part 2), there will be no randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1, Dose Optimization, Cohort 1 (Experimental): HER2-positive or HER2-low, unresectable or metastatic BC.
  Interventions: Drug: BB-1701
- Part 1, Dose Optimization, Cohort 2 (Experimental): HER2-positive or HER2-low, unresectable or metastatic BC.
  Interventions: Drug: BB-1701
- Part 1, Dose Optimization, Cohort 3 (Experimental): HER2-positive or HER2-low, unresectable or metastatic BC.
  Interventions: Drug: BB-1701
- Part 2, Dose Expansion (Experimental): HER2-positive or HER2-low, unresectable or metastatic BC.
  Interventions: Drug: BB-1701

INTERVENTIONS:
Drug: BB-1701 — BB-1701 will be administered as an intravenous infusion, every 3 weeks (21-day cycle).

SUMMARY:
The primary purpose of the Dose Optimization (Part 1) of this study is to assess the safety and tolerability of BB-1701 and to determine the recommended dose (RD) of BB-1701 for Dose Expansion (Part 2). The primary purpose of Dose Expansion (Part 2) is to assess the antitumor activity of BB-1701 at RD in the selected population(s) of breast cancer (BC).

ELIGIBILITY:
Inclusion Criteria

* Male or female, aged >=18 years at the time of informed consent.
* Metastatic or unresectable BC that is histologically confirmed to be either HER2-positive (defined as an immunohistochemistry [IHC] status of 3+, or a positive in situ hybridization [ISH] test [fluorescence, chromogenic, or silver-enhanced ISH] if IHC status is 2+) or HER2-low (defined as an IHC status of 1+, or 2+ and negative ISH) per the American Society of Clinical Oncology/College of American Pathology guidelines as documented prior to trastuzumab deruxtecan (T-DXd) treatment.
* Must have previously received T-DXd.
* Sufficient tumor tissue is required for HER2 status testing at a central laboratory.
* Measurable disease per RECIST 1.1 as assessed by the investigator. Participants with bone only disease may be eligible if there is a measurable soft tissue component associated with the bone lesion.
* Must have previously received at least 1 but no more than 3 prior chemotherapy-based regimes in the unresectable or metastatic setting. If recurrence occurred during or within 6 months of (neo) adjuvant chemotherapy, this would count as 1 line of chemotherapy.
* If HR-positive HER2-low BC, must have previously received endocrine therapy and is not expected to further benefit from it.
* ECOG PS 0 or 1.
* Life expectancy of at least 3 months.
* Adequate organ function and laboratory parameters.

Exclusion Criteria

* Presence of brain or subdural metastases, unless participant has completed local therapy and has discontinued the use of corticosteroids for this indication for at least 2 weeks prior to starting treatment in this study.
* Diagnosed with meningeal carcinomatosis.
* Received anticancer therapy (chemotherapy or other systemic anticancer therapies, immunotherapy, radiation therapy, etc) or an investigational drug or device within the past 28 days or 5 half-lives, whichever is shorter.
* Prior treatment with eribulin.
* Any prior allergic reactions of Grade >=3 to monoclonal antibodies or contraindication to the receipt of corticosteroids or any of the excipients (investigators should refer to the prescribing information for the selected corticosteroid).
* Residual toxic effects of prior therapies or surgical procedures that is Grade >=2 (except alopecia or anemia).
* Grade >=2 peripheral neuropathy or history of Grade >=3 peripheral neuropathy or discontinued any prior treatment due to peripheral neuropathy.
* Active pneumonitis/interstitial lung disease (ILD) or any clinically significant lung disease (example, chronic obstructive pulmonary disease), history of Grade >=2 pneumonitis/ILD, or received radiotherapy to lung fields within 12 months of Cycle 1 Day 1 of study treatment.
* Congestive heart failure greater than (>) New York Heart Association Class II or left ventricular ejection fraction (LVEF) less than (<) 50 percent (%) measured by multigated acquisition scan (MUGA) or echocardiogram.
* Has a corrected QT interval prolongation per Fridericia formula (QTcF) >470 millisecond (ms) (for both males and females) based on screening triplicate 12-lead ECG.
* Concomitant active infection requiring systemic treatment, except:

  * If known to be human immunodeficiency virus (HIV)-positive, must be on anti-HIV therapy for at least 4 weeks and have a clusters of differentiation 4+ T-cell (CD4+) count >=350 cells per microliter (cells/mcL) and an HIV viral load <400 copies per milliliter (copies/mL).
  * If meets the criteria for anti-hepatitis B virus (HBV) therapy, must agree to take anti-HBV therapy, if known to be HBV-positive as defined by positive hepatitis B surface antigen or hepatitis B core antibody. HBV viral load must be undetectable.
  * If known to be hepatitis C virus (HCV)-positive must have completed curative therapy for HCV. HCV viral load must be undetectable.
* Known history of active bacillus tuberculosis (TB).
* Any medical or other condition which, in the opinion of the investigator would preclude the participant's participation in the clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2024-04-10 (Actual); Primary Completion 2025-02-05 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Part 1, Dose Optimization: Number of Participants With Adverse Events (AEs) | Baseline up to 35 months
  An AE is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of an investigational product, whether or not considered related to the investigational product; Any new disease or exacerbation of an existing disease; any deterioration in non-protocol-required measurements of a laboratory value or other clinical test (example, electrocardiogram [ECG] or x-ray) that results in symptoms, a change in treatment, or discontinuation of study drug; Recurrence of an intermittent medical condition (example, headache) not present pretreatment (baseline); An abnormal laboratory test result should be considered an AE if the identified laboratory abnormality leads to any type of intervention, withdrawal of study drug, or withholding of study drug, whether prescribed in the protocol or not. An AE does not necessarily have a causal relationship with the medicinal product.
Part 1, Dose Optimization: Number of Participants With Clinically Significant Laboratory Values | Baseline up to 35 months
  Clinical laboratory parameters includes hematology, chemistry, and urinalysis.
Part 1, Dose Optimization: Number of Participants With Clinically Significant Vital Sign Values | Baseline up to 35 months
  Vital sign parameters includes systolic and diastolic blood pressure (BP), pulse, respiratory rate, body temperature.
Part 1, Dose Optimization: Number of Participants With Clinically Significant 12-lead ECGs Values | Baseline up to 35 months
  Number of participants with clinically significant 12-lead ECGs values will be reported.
Part 1, Dose Optimization: Number of Participants With Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) | Baseline up to 35 months
  Number of participants with ECOG PS will be reported.
Part 1, Dose Optimization: Objective Response Rate (ORR) | From date of first dose of study drug until first documentation of CR or PR (up to 35 months)
  ORR is defined as the percentage of participants achieving a confirmed complete response (CR) or confirmed partial response (PR) by investigator assessment per Response Evaluation Criteria for Solid Tumours (RECIST) version (v) 1.1.
Part 2, Dose Expansion: Objective Response Rate (ORR) Based on Blinded Independent Central Review (BICR) Assessment per RECIST v1.1 | From date of first dose of study drug until first documentation of CR or PR (up to 35 months)
  ORR is defined as the percentage of participants achieving a confirmed CR or confirmed PR based on BICR assessment per RECIST v1.1.

SECONDARY OUTCOMES:
Part 1, Dose Optimization: Duration of Response (DOR) | From the date of documented CR or PR to the date of PD or death, whichever occurs first (up to 35 months)
  DOR defined as the time from the onset date of documented CR or PR for confirmed responses by investigator per RECIST v1.1 to the date of disease progression (PD) or death, whichever occurs first.
Part 1, Dose Optimization: Progression-free Survival (PFS) | From the date of first dose to the date of the first documentation of PD or death, whichever occurs first (up to 35 months)
  PFS is defined as the time from the date of first dose to the date of the first documentation of PD by investigator per RECIST v1.1 or death, whichever occurs first.
Part 1, Dose Optimization: Overall Survival (OS) | From the date of first dose to the date of death (up to 35 months)
  Overall survival (OS) is defined as the time from the date of first dose to the date of death. OS will be based on Kaplan-Meier estimates.
Part 1, Dose Optimization: Disease Control Rate (DCR) | From the date of first dose until PD or death, whichever occurs first (up to 35 months)
  DCR is defined as the percentage of participants with CR, PR, or stable disease (SD) (greater than or equal to [>=] 5 weeks from the first dose) by investigator per RECIST v1.1.
Part 1, Dose Optimization: Clinical Benefit Rate (CBR) | From the date of first dose until PD or death, whichever occurs first (up to 35 months)
  CBR is defined as the percentage of participants with CR, PR, or durable SD (duration of SD >=23 weeks) by investigator per RECIST v1.1.
Part 1, Dose Optimization: Time to Response (TTR) | From the date of first dose to the day of the first documented CR or PR (up to 35 months)
  TTR is defined as the time from the date of first dose to the day of the first documented CR or PR for confirmed responses by investigator per RECIST v1.1
Part 1, Dose Optimization, Cmax: Maximum Observed Concentration of BB-1701, Total Antibody and Eribulin (Payload) | Baseline up to 35 months
Part 1, Dose Optimization, Tmax: Time to Reach Maximum Observed Concentration (Cmax) of BB-1701, Total Antibody and Eribulin (Payload) | Baseline up to 35 months
Part 1, Dose Optimization, AUC(0-t): Area Under the Concentration-time Curve From Zero Time to Time of Last Quantifiable Concentration of BB-1701, Total Antibody and Eribulin (Payload) | Baseline up to 35 months
Part 1, Dose Optimization, AUC(0-inf): Area Under the Concentration-time Curve From Zero Time to Infinity of BB-1701, Total Antibody and Eribulin (Payload) | Baseline up to 35 months
Part 1, Dose Optimization, t1/2: Terminal Phase Elimination Half-life of BB-1701 | Baseline up to 35 months
Part 1, Dose Optimization, CL: Total Body Clearance of BB-1701 | Baseline up to 35 months
Part 1, Dose Optimization, Vss: Volume of Distribution at Steady State for BB-1701 | Baseline up to 35 months
Part 1, Dose Optimization, Ctrough: Trough Concentration of BB-1701 | Baseline up to 35 months
Part 1, Dose Optimization: Statistical Correlation Between Serum Concentrations of BB-1701 with ORR and AEs | Baseline up to 35 months
Part 2, Dose Expansion: Duration of Response (DOR) Based on BICR Assessment by RECIST v1.1 | From the date of documented CR or PR to the date of PD or death, whichever occurs first (up to 35 months)
  DOR is defined as the time from the onset date of documented CR or PR for confirmed responses based on BICR by RECIST v1.1 to the date of PD or death, whichever occurs first.
Part 2, Dose Expansion: Disease Control Rate (DCR) Based on BICR Assessment per RECIST v1.1 | From the date of first dose until first documentation of CR or PR or SD (up to 35 months)
  DCR is defined as the percentage of participants with CR, PR, or stable disease (SD) (>=5 weeks from the first dose) based on BICR per RECIST v1.1.
Part 2, Dose Expansion: Time to Response (TTR) Based on BICR Assessment per RECIST v1.1 | From the date of first dose to the day of the first documented CR or PR (up to 35 months)
  TTR is defined as the time from the date of first dose to the day of the first documented CR or PR for confirmed responses based on BICR per RECIST v1.1
Part 2, Dose Expansion: Clinical Benefit Rate (CBR) Based on BICR Assessment per RECIST v1.1 | From the date of first dose until PD or death, whichever occurs first (up to 35 months)
  CBR is defined as the percentage of participants with CR, PR, or durable SD (duration of SD >=23 weeks) based on BICR per RECIST v1.1.
Part 2, Dose Expansion: Progression-free Survival (PFS) Based on BICR Assessment per RECIST v1.1 | From the date of first dose to the date of the first documentation of PD or death, whichever occurs first (up to 35 months)
  PFS is defined as the time from the date of first dose to the date of the first documentation of PD based on BICR per RECIST v1.1 or death, whichever occurs first.
Part 2, Dose Expansion: Overall Survival (OS) | From the date of first dose to the date of death (up to 35 months)
  Overall survival (OS) is defined as the time from the date of first dose to the date of death. OS will be based on Kaplan-Meier estimates.
Part 2, Dose Expansion: Number of Participants With AEs | Baseline up to 35 months
  An AE is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of an investigational product, whether or not considered related to the investigational product; Any new disease or exacerbation of an existing disease; any deterioration in non-protocol-required measurements of a laboratory value or other clinical test (example, ECG or x-ray) that results in symptoms, a change in treatment, or discontinuation of study drug; Recurrence of an intermittent medical condition (example, headache) not present pretreatment (baseline); An abnormal laboratory test result should be considered an AE if the identified laboratory abnormality leads to any type of intervention, withdrawal of study drug, or withholding of study drug, whether prescribed in the protocol or not. An AE does not necessarily have a causal relationship with the medicinal product.
Part 2, Dose Expansion: Number of Participants With Clinically Significant Laboratory Values | Baseline up to 35 months
  Clinical laboratory parameters includes hematology, chemistry, and urinalysis.
Part 2, Dose Expansion: Number of Participants With Clinically Significant Vital Sign Values | Baseline up to 35 months
  Vital sign parameters includes systolic and diastolic BP, pulse, respiratory rate, body temperature.
Part 2, Dose Expansion: Number of Participants With Clinically Significant 12-lead ECGs Values | Baseline up to 35 months
  Number of participants with clinically significant 12-lead ECGs values will be reported.
Part 2, Dose Expansion: Number of Participants With Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) | Baseline up to 35 months
  Number of participants with ECOG PS will be reported.

CONTACTS AND LOCATIONS:
Locations (49):
- United States (27):
  - Cancer and Blood Specialty Clinic, Los Alamitos, California
  - UCLA Center for East-West Medicine, Los Angeles, California
  - UCSF, San Francisco, California
  - Yale New Haven Hospital, New Haven, Connecticut
  - AdventHealth Cancer Institute - Orlando, Orlando, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Fort Wayne Medical Oncology & Hematology, Fort Wayne, Indiana
  - Community Cancer Center South, Indianapolis, Indiana
  - Mission Blood and Cancer, Des Moines, Iowa
  - University of Michigan Hospital, Ann Arbor, Michigan
  - Washington University in St. Louis School of Medicine, St Louis, Missouri
  - NHO Revive Research Institute LLC, Lincoln, Nebraska
  - Nebraska Cancer Specialist, Omaha, Nebraska
  - Astera Cancer Care, East Brunswick, New Jersey
  - Summit Medical Group, Florham Park, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - New Mexico Oncology Hematology Consultants, Albuquerque, New Mexico
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Cleveland Clinic - Fairview Hospital - Cancer Center (Moll Cancer Center), Cleveland, Ohio
  - Cleveland Clinic - Hillcrest Hospital - Hillcrest Cancer Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Oncology Specialists, Salem, Oregon
  - UPMC CancerCenter at Magee - Womens Hospital, Pittsburgh, Pennsylvania
  - St. Francis Cancer Center, Greenville, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - The West Clinic, PLLC dba West Cancer Cente, Germantown, Tennessee
  - Northwest Medical Specialties, Puyallup, Washington
- France (4):
  - CHU Besançon - Hôpital Jean Minjoz, Besançon
  - Institut Régional du Cancer de Montpellier, Montpellier
  - Centre Armoricain de Radiotherapie Imagerie & Oncologie (CARIO), Plérin
  - Institut de Cancerologie de Ouest (ICO) - Saint-Herblain, Saint-Herblain
- Japan (15):
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Hiroshima City Hiroshima Citizens Hospital, Hiroshima, Hiroshima
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Hyogo Medical University Hospital, Nishinomiya-shi, Hyōgo
  - Sagara Hospital, Social Medical Corporation Hakuaikai, Kagoshima, Kagoshima-ken
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - National Cancer Center Hospital (NCCH), Chūōku, Kansai
  - Kyoto University Hospital, Sakyo-ku, Kyoto
  - Tohoku University Hospital, Sendai, Miyagi
  - Okayama University Hospital, Okayama, Okayama-ken
  - Saitama Medical University International Medical Center, Hidaka-shi, Saitama
  - Saitama Cancer Center, Kitaadachi-gun, Saitama
  - St. Luke's International Hospital, Chuou-ku, Tokyo
  - The Cancer Institute Hospital of Japanese Foundation for Cancer Research, Koto Ku, Tokyo
  - Showa University, Shinagawa Ku, Tokyo
- Spain (3):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - HM Universitario Sanchinarro, Madrid
  - Hospital Beata María Ana, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.